CLINICAL TRIAL: NCT02226549
Title: A Phase 2, Randomized, Open-Label Study of Ledipasvir/Sofosbuvir Fixed-Dose Combination and Vedroprevir With or Without Ribavirin in Treatment-Experienced Subjects With Chronic Genotype 1 HCV Infection and Cirrhosis
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination and Vedroprevir With or Without Ribavirin in Treatment-Experienced Participants With Chronic Genotype 1 HCV Infection and Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1512
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2016-02

CONDITIONS: Hepatitis C Virus Infection
Keywords: hepatitis C; Gilead; GS-9451
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination; GS-9451

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDV/SOF+VDV (Experimental): Participants will receive LDV/SOF+VDV for 8 weeks.
  Interventions: Drug: LDV/SOF; Drug: VDV
- LDV/SOF+VDV+RBV (Experimental): Participants will receive LDV/SOF+VDV+RBV for 8 weeks.
  Interventions: Drug: LDV/SOF; Drug: VDV; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — LDV/SOF (90/400 mg) FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: VDV — VDV 80 mg tablet administered orally once daily
  Other Names: GS-9451
Drug: RBV — RBV tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF+VDV+RBV

SUMMARY:
This study is to evaluate the antiviral efficacy, safety, and tolerability of combination therapy with ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) + vedroprevir (VDV) ± ribavirin (RBV) for 8 weeks in treatment-experienced adults with chronic genotype 1 hepatitis C virus (HCV) infection and cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, with chronic HCV genotype 1 infection
* Documentation as treatment-experienced having received pegylated interferon (Peg-IFN) + RBV ≥ 4 weeks of duration without an additional agent in the regimen without achieving sustained viral response (SVR)
* Presence of compensated cirrhosis
* Screening laboratory values within defined thresholds
* Must use specific contraceptive methods if female of childbearing potential or sexually active male
* Not pregnant or a nursing female

Exclusion Criteria:

* Co-infection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hyland, DPhil, Study Director — Gilead Sciences
Locations (1):
- San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 study site in the United States. The first participant was screened on 24 July 2014. The last study visit occurred on 06 February 2015.
Pre-assignment Details: 72 participants were screened.
Groups:
- LDV/SOF+VDV: Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet + vedroprevir (VDV) 80 mg tablet once daily for 8 weeks
- LDV/SOF+VDV+RBV: LDV/SOF (90/400 mg) FDC tablet once daily + VDV 80 mg tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 8 weeks
Period: Overall Study
Arm/Group | LDV/SOF+VDV | LDV/SOF+VDV+RBV
Started | 23 | 24
Completed | 22 | 23
Not Completed | 1 | 1
Not completed — Randomized but Never Treated | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug.
Groups:
- LDV/SOF+VDV: LDV/SOF (90/400 mg) FDC tablet + VDV 80 mg tablet once daily for 8 weeks
- LDV/SOF+VDV+RBV: LDV/SOF (90/400 mg) FDC tablet once daily + VDV 80 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 8 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF+VDV | LDV/SOF+VDV+RBV | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (7.9) | 56 (7.7) | 57 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 12 | 18 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 1 | 2
  White | 21 | 23 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 6 | 11 | 17
  Not Hispanic or Latino | 16 | 12 | 28
  Not Permitted | 0 | 1 | 1
HCV Genotype [Number; unit: participants]
  Genotype 1a | 14 | 18 | 32
  Genotype 1b | 7 | 6 | 13
  Genotype 1a,1b | 1 | 0 | 1
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 4 | 1 | 5
    CT | 12 | 16 | 28
    TT | 6 | 6 | 12
    Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+VDV | LDV/SOF+VDV+RBV
Number analyzed (Participants) | 22 | 24
percentage of participants | 95.5 | 87.5

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 8 weeks
Population: Safety Analysis Set: participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+VDV | LDV/SOF+VDV+RBV
Number analyzed (Participants) | 22 | 24
percentage of participants | 0 | 8.3

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+VDV | LDV/SOF+VDV+RBV
Number analyzed (Participants) | 22 | 24
percentage of participants | 95.5 | 95.8

ADVERSE EVENTS:
Time Frame: Up to 8 weeks plus 30 days
Description: Safety Analysis Set: participants who received at least 1 dose of study drug.
Arm/Group | LDV/SOF+VDV | LDV/SOF+VDV+RBV
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 7/22 | 12/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF+VDV (N=22) | LDV/SOF+VDV+RBV (N=24)
Fatigue (General disorders) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 3
Headache (Nervous system disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years